CLINICAL TRIAL: NCT04733248
Title: Effectiveness of Kinesiotaping on Patient's Functional Status in Non-specific Neck Pain
Brief Title: kINESIOTAPING ON PATIENT'S FUNCTIONAL STATUS IN NON-SPECIFIC NECK PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Assistant professor, Aqua Medical Services (Pvt) Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aneeqa Gull 00378
Record Dates: First submitted 2020-12-22; First posted 2021-02-02 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Neck Pain
Keywords: Superficial Back Muscles; Exercise Therapy; Physical Therapy Modalities; Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping group (Active Comparator): Hot pack, Tens, stretching exercises, Kinesiotaping (I-O) and Home plan
  Interventions: Other: Kinesiotaping group
- stretching group (Experimental): Hot pack, Tens, stretching exercises and Home plan
  Interventions: Other: stretching group

INTERVENTIONS:
Other: Kinesiotaping group — * HOT PACK (10 MINTS)
  * TENS(10 MINTS)
  * STRETCHING EXERCISES(10 reps 3sets) hold for 2 sec
  * Apply KINESO- TAPE on upper trapezius (from I-O for Inhibition purpose)
  HOME PLAN OF EXPERIMENTAL GROUP:
  * SELF STRECHINGS (10 reps 3 sets)
  * AROMS
  * NECK ISOMETRICS (10 reps 3 sets)hold for 10 sec (In neck flexion, In neck extension, In side bending) In experimental group kinesiotape was applied on upper trapezius from insertion to origin for inhibition purpose. As it had increased the functional status of the patient. Post -intervention assessment was taken on 1 st, 2nd and 3rd visit.
  Arms: Kinesiotaping group
Other: stretching group — * HOT PACK (10 MINTS)
  * TENS(10 MINTS)
  * STRETCHINGS EXERCISES (10 reps 3sets) hold for 2 sec 5.9HOME PLAN OF CONTROL GROUP:
  * SELF STRECHINGS (10 reps 3 sets)
  * AROMS
  * NECK ISOMETRICS (10 reps 3 sets)hold for 10 sec In neck flexion In neck extension In side bending Post-intervention assessment was taken on 1 st, 2nd and 3 rd visit
  Arms: stretching group

SUMMARY:
The objective of the study is to find the effectiveness of kinesiotaping on the patient's functional status in non-specific neck pain. This is an RCT in which 26 participants with non-specific neck pain who fulfilled the inclusion criteria were included in the study. Individuals were randomly allocated into two groups (control and experimental) by using a sealed envelope method. The treatment protocol given to the experimental group includes kinesiotaping on upper trapezius muscle using inhibition technique (I-O) along with exercise therapy while in the control group exercise therapy was given alone. Data was collected by using NPRS and NDI. Pre and post assessment was taken on 1 st, 2nd, and 3rd sessions, and each session was 3 days apart. Parametric tests including independent T-test and paired T-test were applied for analyzing normal data. while non-parametric tests including Mann Whitney and Wilcoxon were applied for nonnormal data analysis.

DETAILED DESCRIPTION:
As expected, the prevalence increases with longer prevalence periods, and generally, women have more NP than men. Neck pain (NP) is a major public health problem, both in terms of personal health and overall well-being as well as indirect expense. For instance, the total cost of NP in the Netherlands in 1996 was estimated at about 1% of the total health care expenditure or 0.1% of the Dutch gross domestic product.Accurate prevalence estimates are desirable to serve as a basis for etiological studies and health care evaluation, and to assess the effect of NP in general populations. Unfortunately, prevalence studies on NP show great variation in both quality and results. For instance, the point prevalence varies between 6% and 22%, and 1-year prevalence between 1.5% and 75%.Neck pain is becoming increasingly common throughout the world. It has a considerable impact on individuals and their families, communities, health-care systems, and businesses. The estimated 1-year incidence of neck pain from available studies ranges between 10.4% and 21.3% with a higher incidence noted in office and computer workers. While some studies report that between 33% and 65% of people have recovered from an episode of neck pain at 1 year, most cases run an episodic course over a person's lifetime, and, thus, relapses are common. The overall prevalence of neck pain in the general population ranges between 0.4% and 86.8% (mean: 23.1%); point prevalence ranges from 0.4% to 41.5% (mean: 14.4%); and 1 year prevalence ranges from 4.8% to 79.5% (mean: 25.8%). Prevalence is generally higher in women, higher in high-income countries compared with low- and middle-income countries, and higher in urban areas compared with rural areas. Many environmental and personal factors influence the onset and course of neck pain. Most studies indicate a higher incidence of neck pain among women and an increased risk of developing neck pain until the 35-49-year age group, after which the risk begins to decline. The Global Burden of Disease 2005 Study is currently making estimates of the global burden of neck pain in relation to impairment and activity limitation, and results will be available in 2011. Nonspecific or simple neck pain, is the most common form of pain in the neck, affecting two out of three people at some point in their lives. While the exact etiology of the pain is often unknown, most cases of non-specific neck pain are caused by mechanical factors such as sprains and strains of the muscles or ligaments in the neck. Inflammation of the facet joints or the joints between the vertebrae leads to an aggravation of these structures during movement (i.e. when turning or bending the neck), giving rise to pain.Other factors that can contribute to the development of mechanical neck pain include Poor posture (i.e. prolonged sitting in a 'bent-forward' position), Physical overload, Stress, Smoking, and Poor psychological health, etc.Most cases of nonspecific neck pain are acute and resolve within three to six weeks with minimal intervention, although some people suffer from recurrent pain. However, if neck pain persists for longer than three months, it is considered chronic and further treatment may be warranted. Furthermore, if neck pain persists or gets worse, it can cause numbness or referral pain in the arm.In general, neck pain refers to pain that occurs between the occipital bone, thoracic vertebra, and shoulder joint. While the majority of people suffer from non-specific or mechanical neck pain, other types of neck pain.Symptoms of non-specific neck pain include Stiff neck, Restricted movement of the neck, Pain when moving the neck, which may spread down an arm and even into the finger, Sensation of 'pins and needles' in part of an arm or hand (caused by irritation of a nerve from the neck/spinal cord going to the arm), Crunching sound when bending or turning the neck.The Kinesio Taping Method is a definitive rehabilitative taping technique that is designed to facilitate the body's natural healing process while providing support and stability to muscles and joints without restricting the body's range of motion as well as providing extended soft tissue manipulation to prolong the benefits of manual therapy administered within the clinical setting. Latex-free and wearable for days at a time, Kinesio Tex Tape is safe for populations ranging from pediatric to geriatric, and successfully treats a variety of orthopedic, neuromuscular, neurological, and other medical conditions. The Kinesio Taping Method is a therapeutic taping technique not only offering patients the support they are looking for, but also rehabilitating the affected condition as well. By targeting different receptors within the somatosensory system, Kinesio Tex Tape alleviates pain and facilitates lymphatic drainage by microscopically lifting the skin. This lifting affect forms convolutions in the skin thus increasing interstitial space and allowing for a decrease in inflammation of the affected areas.Based upon years of clinical use, Kinesio Tex Tape is specifically applied to the patient based upon their needs after evaluation. The findings of the clinical evaluation or assessment dictate the specifics of the Kinesio Tex Tape application and other possible treatments or modalities. With the utilization of single "I" strips or modifications in the shape of an "X", "Y" or other specialized shapes as well as the direction and amount of stretch placed on the tape at the time of application, Kinesio Tex Tape can be applied in hundreds of ways and has the ability to re-educate the neuromuscular system, reduce pain and inflammation, optimize performance, prevent injury and promote good circulation and healing, and assist in returning the body to homeostasis.Evaluation and assessment are key to the treatment of any clinical condition. In order to get the desired results from a Kinesio Tex Tape application as well as any other treatment, a full assessment of the patient is necessary. In some cases, the treatment of a condition may require treatment of other underlying conditions as well. This assessment should include manual muscle testing, range of motion testing, gait assessment, and any other orthopedic special tests that you deem necessary. The information gained from these assessments will allow for the proper treatment protocol to be laid out. Kinesio Tex Tape can be a valuable addition to this protocol. It has been proven to have positive physiological effects on the skin, lymphatic and circulatory system, fascia, muscles, ligaments, tendons, and joints. It can be used in conjunction with a multitude of other treatments and modalities within the clinic and is effective during the rehabilitative and chronic phases of an injury as well as being used for preventative measures.It includes surgical versus non-surgical treatment options.Neck pain is a common complaint. Many Conservative treatments are available to patients and accepted as standard forms of practice, including such common conservative strategies as medication, physical medicine methods, manual treatments, and education of patients.The best advice for recovering from simple neck pain is to use anti-inflammatory medications or muscle relaxants to ease the pain and to resume normal activities as soon as possible. Gently moving the neck in all directions several times a day will prevent the neck from stiffening up.Treatment options for mechanical neck pain include Physiotherapy (i.e. heat, cold, traction, manipulation), Gentle neck exercises, Learning proper sitting posture, Yoga for improving neck posture, Massage therapy, Pressure point therapy, and Kinesio taping. Kinesiology taping (KT) is a therapeutic tool and has become increasingly popular within the sporting arena. Taping has been used for a long time for the prevention and treatment of sporting injuries. KT is not only used for sporting injuries but for a variety of other conditions. It was developed by Japanese chiropractor Kenzo Kase in the 1970s with the intention to alleviate pain and improve the healing in soft tissues. There are many proposed benefits to KT, including proprioceptive facilitation; reduced muscle fatigue; muscle facilitation; reduced delayed-onset muscle soreness; pain inhibition; enhanced healing, such as reducing edema, and improvement of lymphatic drainage and blood flow.An RCT was conducted which concluded that In daily practice, manual therapy is a favorable treatment option for patients with neck pain compared with physical therapy or continued care by a general practitioner. Patients with acute WAD receiving an application of Kinesio Taping, applied with proper tension, exhibited statistically significant improvements immediately following application of the Kinesio Tape and at a 24-hour follow-up. However, the improvements in pain and cervical range of motion were small and may not be clinically meaningful. Future studies should investigate if Kinesio Taping provides enhanced outcomes when added to physical therapy interventions with proven efficacy or when applied over a longer period. Patients with mechanical neck pain who received cervical thrust manipulation or Kinesio Taping exhibited similar reductions in neck pain intensity and disability and similar changes in active cervical range of motion, except for rotation. Changes in neck pain surpassed the minimal clinically important difference, whereas changes in disability did not. Changes in cervical range of motion were small and not clinically meaningful. Because investigators did not include a control or placebo group in this study, investigators cannot rule out a placebo effect or natural changes over time as potential reasons for the improvements measured in both groups. This study shows that Kinesio Taping leads to improvements in pain, pressure pain threshold, and cervical range of motion, but not a disability in a short time. Therefore, Kinesio Taping can be used as an alternative therapy method in the treatment of patients with MPS.

ELIGIBILITY:
Inclusion Criteria:

* Age b/w 25-55 years
* Limited ROM
* Pain more than 3on NPRS
* Individuals having NDI score 15 - 24 = moderate,25-34 = severe

Exclusion Criteria:

* Radiculopathies
* Malignancy
* infection
* trauma

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
numeric pain rating scale | 2 weeks
  It is numeric pain rating scale for measuring pain intensity. it ranges from 0-10.In which 0 shows no pain,1-3 (mild pain),4-6(moderate pain) and 10 shows severe pain. As guided by the researcher, pain intensity was marked by the patient

SECONDARY OUTCOMES:
neck disability index scale | 2 weeks
  It is the neck disability index scale and was first developed in 1989 by HowardVernon. it is standard for measuring neck disability due to neck pain. This scale includes 10 items. Each of 10 items score from 0-5.Maximum score is 50.In which 0-4 shows no disability,5-14 shows mild disability level,15-24 presents moderate level of disability,25-34 shows severe disability level while >34 predicts complete disability. It is used by the clinician to determine patient's functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad,, PHD*, Principal Investigator — Shifa Tameer e milat University
Locations (1):
- Aqua research Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] McLean SM, May S, Klaber-Moffett J, Sharp DM, Gardiner E. Risk factors for the onset of non-specific neck pain: a systematic review. J Epidemiol Community Health. 2010 Jul;64(7):565-72. doi: 10.1136/jech.2009.090720. Epub 2010 May 12. PMID 20466711
- [Background] Auvinen JP, Tammelin TH, Taimela SP, Zitting PJ, Jarvelin MR, Taanila AM, Karppinen JI. Is insufficient quantity and quality of sleep a risk factor for neck, shoulder and low back pain? A longitudinal study among adolescents. Eur Spine J. 2010 Apr;19(4):641-9. doi: 10.1007/s00586-009-1215-2. Epub 2009 Nov 20. PMID 19936804
- [Background] Castro-Sanchez AM, Lara-Palomo IC, Mataran-Penarrocha GA, Fernandez-Sanchez M, Sanchez-Labraca N, Arroyo-Morales M. Kinesio Taping reduces disability and pain slightly in chronic non-specific low back pain: a randomised trial. J Physiother. 2012;58(2):89-95. doi: 10.1016/S1836-9553(12)70088-7. PMID 22613238
- [Background] Lim EC, Tay MG. Kinesio taping in musculoskeletal pain and disability that lasts for more than 4 weeks: is it time to peel off the tape and throw it out with the sweat? A systematic review with meta-analysis focused on pain and also methods of tape application. Br J Sports Med. 2015 Dec;49(24):1558-66. doi: 10.1136/bjsports-2014-094151. Epub 2015 Jan 16. PMID 25595290
- [Background] Kachanathu SJ, Alenazi AM, Seif HE, Hafez AR, Alroumim MA. Comparison between Kinesio Taping and a Traditional Physical Therapy Program in Treatment of Nonspecific Low Back Pain. J Phys Ther Sci. 2014 Aug;26(8):1185-8. doi: 10.1589/jpts.26.1185. Epub 2014 Aug 30. PMID 25202177
- [Background] Shih HS, Chen SS, Cheng SC, Chang HW, Wu PR, Yang JS, Lee YS, Tsou JY. Effects of Kinesio taping and exercise on forward head posture. J Back Musculoskelet Rehabil. 2017;30(4):725-733. doi: 10.3233/BMR-150346. PMID 28282792
- [Background] Pelosin E, Avanzino L, Marchese R, Stramesi P, Bilanci M, Trompetto C, Abbruzzese G. kinesiotaping reduces pain and modulates sensory function in patients with focal dystonia: a randomized crossover pilot study. Neurorehabil Neural Repair. 2013 Oct;27(8):722-31. doi: 10.1177/1545968313491010. Epub 2013 Jun 13. PMID 23764884
- [Background] Hurwitz EL, Carragee EJ, van der Velde G, Carroll LJ, Nordin M, Guzman J, Peloso PM, Holm LW, Cote P, Hogg-Johnson S, Cassidy JD, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Treatment of neck pain: noninvasive interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S123-52. doi: 10.1097/BRS.0b013e3181644b1d. PMID 18204386